CLINICAL TRIAL: NCT04642560
Title: Compliance With AntibIotic TherapY Guidelines in French Pediatric Intensive Care Units
Brief Title: Compliance With AntibIotic TherapY Guidelines in French PICUs
Acronym: COMITY
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0416
Record Dates: First submitted 2020-07-29; First posted 2020-11-24 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Bacterial Infections
Keywords: Children; Pediatric Intensive Care Unit; Antibiotic duration; Compliance; Guidelines
MeSH Terms: conditions — Bacterial Infections; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Usual practice: Any child hospitalized in Pediatric or Neonatal ICU and receiving systemic (intravascular, intramuscular or oral) antibiotic treatment for an episode of suspected or proven community-acquired or nosocomial bacterial infection

SUMMARY:
This observational, prospective, multicenter study, conducted in nine French Pediatric and Neonatal Intensive Care Units (ICUs), will assess the antibiotic therapy for a child hospitalized in ICU and receiving systemic antibiotics for an episode of suspected or proven community-acquired or nosocomial bacterial infection. The study will describe the mean duration of antibiotic therapy, as well as compliance with the recommendations concerning the duration of antibiotic therapy, the choice of antibiotics, the daily dosage and the number of doses per 24 hours according to the type of bacterial infection. Patients will be monitored until the end of their hospitalization.

DETAILED DESCRIPTION:
Bacterial infections are widespread in Pediatric and Neonatal ICU, and antibiotic treatments are widely used. The Surviving Sepsis Campaign (SSC) recommends the early administration of empiric broad-spectrum antibiotic therapy in the event of suspected bacterial infection, with de-escalation once the pathogen is identified and sensitivities established. Standard-of-care of antibiotic treatment and duration is determined by the type of infection, microbiological results, and clinical biological evolution (improvement is demonstrated by reduction of fever, pain, and local signs as well as a decrease of the biological inflammatory syndrome [leukocyte count, C-reactive protein]) and/or radiological evolution, according to published guidelines: French guidelines (Société de Pathologie Infectieuse de Langue Française [SPILF], Groupe de Pathologies Infectieuses en Pédiatrie [GPIP], Société Française d'Anesthésie et de Réanimation [SFAR], Société de Réanimation de Langue Française [SRLF], Haute Autorité de Santé [HAS]), European guidelines (European Society of Clinical Microbiology and Infectious Diseases [ESCMID]), American guidelines (Infectious Diseases Society of America [IDSA], American Society of Clinical Oncology [ASCO]), and Australian guidelines (Australasian Society for Infectious Diseases). These recommendations are numerous. Compliance with these recommendations has never been evaluated in Pediatric and Neonatal ICU. Long courses of antibiotic treatment increase the duration of hospitalization and are associated with changes in the microbiome, emergence of multidrug resistant organisms, and antibiotic-associated adverse events (toxicity, overdose, allergy). On the other hand, too short antibiotic therapy can expose the patient to a risk of infection recurrence.

The 2020 SSC pediatric guidelines identified the use of procalcitonin to guide antimicrobial therapy and its relationship to patients' outcome as a future research opportunity. However, in order to demonstrate a decrease in the antibiotic course in the PCT-guided antibiotic therapy group compared with the standard-of-care antibiotic therapy group in future interventional studies in critically ill children, calculating the number of subjects required demands knowledge of the mean duration of antibiotic therapy and the standard deviation (SD) in the standard group. These data are unknown in France.

In this context, the study suggest evaluating the mean duration of antibiotic therapy for a child hospitalized in a French Pediatric and Neonatal ICU and receiving systemic antibiotics for an episode of suspected or proven community-acquired or nosocomial bacterial infection, as well as compliance with recommendations concerning the antibiotic duration, the choice of antibiotics, the daily dose and the number of doses per 24 hours according to the type of bacterial infection.

This is a French observational, prospective, multicenter study in Pediatric and Neonatal ICU. All children hospitalized in Pediatric or Neonatal ICU and receiving systemic (intravascular, intramuscular or oral) antibiotic treatment for a suspected or proven community-acquired or nosocomial bacterial infection are eligible. The day of antibiotic therapy initiation at appropriate doses for the suspected or proven bacterial infection corresponds to day 0 (D0). Detailed information about the bacterial infection type (including origin of the infection [community or nosocomial], initially infection site(s), final diagnosis for the episode [no bacterial infection, presumed bacterial infection, or documented bacterial infection], sepsis severity according to 2005 International Pediatric Sepsis Consensus conference [IPSC], infection site(s) ultimately identified, causative bacteria, multidrug-resistant bacteria, bacteremia, presence or absence of toxinic signs/infected thrombophlebitis/infective endocarditis/secondary localization), acute organ dysfunctions (2005 IPSC, Pediatric Logistic Organ Dysfunction-2 [PELOD-2], and Pediatric Sequential Organ Failure Assessment [pSOFA] scores), antimicrobial, non-infectious associated treatment, and any antibiotics-related adverse effects will be will be prospectively openly recorded by medical study site investigators and reported in a standardized Case Report Form (CRF) every day until cessation of antibiotics in hospital (in ICU and in general department if antibiotic therapy is not completed in the ICU). At the end of hospitalization, a visit will be conducted to collect dates of discharge from the ICU and hospital, patient clinical status on discharge, detailed data from the ambulatory antibiotic therapy for the first episode based on discharge medical prescription (if the patient is discharged from hospital with antibiotic treatment for the first bacterial infection), recurrence of infection occurring in the same hospital stay as for the first episode, detailed antibiotic therapy for infection recurrence according to the patient's medical file for recurrence's antibiotics in hospital and to the medical prescription for recurrence's antibiotics continued in ambulatory care, and any antibiotics-related adverse effects.

For the entire study population, the same pediatric infectious disease expert committee will analyze the gap between treatment and current recommendations (choice of antibiotics, daily dose, number of doses administered per 24 hours and total duration of antibiotic therapy). For each type of infection, the mean duration (SD) of antibiotic treatment administered will be compared with the recommended duration of antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Neonates, infants and children hospitalized in Pediatric or Neonatal ICU and receiving systemic (intravascular, intramuscular or oral) antibiotic treatment for less than 24 hours with appropriate dosages for an episode of suspected or proven community-acquired or nosocomial bacterial infection.
* Informed verbal consent obtained from both parents or legal guardians.

Exclusion Criteria:

* Newborns <72 hours old.
* Neonates <37 weeks of corrected gestational age.
* Age ≥18 years.
* Antibiotic prophylaxis.
* Children previously included in an interventional study in progress.

Ages: 72 Hours to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any child hospitalized in Pediatric or Neonatal ICU and receiving systemic (intravascular, intramuscular or oral) antibiotic treatment for less than 24 hours with appropriate dosages for an episode of suspected or proven community-acquired or nosocomial bacterial infection.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients (%) for whom there is a gap between practices and current recommendations regarding the duration of antibiotic therapy (between beginning of antibiotics and cessation of antibiotics) | up to cessation of antibiotics in hospital up to 3 month
  It includes only the length of treatment for the initial suspected or proven bacterial infection episode but not for recurrences. The duration of antibiotic therapy for the first episode of suspected or proven bacterial infection is the time interval, expressed in days, between the starting time of systemic (intravenous, intramuscular or oral) antibiotics with appropriate dosages (D0) and the stopping time of the antibiotic therapy. Detailed information about antibiotic treatment will be collected every day of hospitalization. If the patient is discharged from hospital with ambulatory antibiotic therapy for the first episode, we will refer to the discharge medical prescription for the complete antimicrobial therapy for the first bacterial infection.

SECONDARY OUTCOMES:
Percentage of patients (%) with recurrence of infection within 28 days following Days 0 | up to 28 days
  The recurrence of infection is defined as the isolation of one or more of the initial causative bacteria from the same or another site at 48 hours or more after cessation of antibiotics, combined with clinical signs or symptoms of infection, or the need to prescribe a new antimicrobial therapy covering this pathogen. Only recurrences treated by antibiotics in the same hospital stay as for the first episode will be taken into account.
Mean (SD) total duration of antibiotic therapy (in days), including the first episode and recurrences within 28 days following D0. | up to 28 days
  The duration of antibiotic therapy for the recurrence of infection is the time interval, expressed in days, between the starting time of a new antimicrobial therapy (intravenous, intramuscular or oral) covering the initial causative bacteria (within 28 days following D0) and the stopping time of this antibiotic therapy (even if it occurs after 28 days following D0). Detailed information about antibiotic treatment for recurrence will be collected on the last day of hospitalization if the patient is discharged from hospital before D28, and on D28 if the patient is discharged from hospital after D28.
Mean (SD) duration of broad-spectrum antibiotic therapy (in days), including the first episode and recurrences within 28 days following D0 | up to 28 days
  Historically, the term "broad-spectrum antibiotics" was used to designate antibiotics that were effective against both gram-positive and gram-negative bacteria. Lately, the World Health Organization have published the 2019 AWaRe classification. It includes 180 antibiotics classified in 3 stewardship groups: Access, Watch and Reserve. We will use separetly both definitions to identify broad-spectrum antibiotics.
  We will not consider the following antibiotics: all antibiotics which have an useful activity against only Gram-positive bacteria (penicillin G, oxacillin, vancomycin, teicoplanin, linezolid, macrolides, clindamycin), and those whose main activity is against Gram-positive bacteria (amoxicillin, 1st generation cephalosporin: cefazolin, cephalexin), 2nd generation cephalosporin (cefuroxim, cefaclor, cefamandol, rifampicin).
  According to the AWaRe classification, we will consider as broad-spectrum antibiotics those from Watch and Reserve groups.
Percentage of patients (%) for whom there is a gap between practices and current recommendations (between beginning of antibiotics and cessation of antibiotics) | up to cessation of antibiotics in hospital
  Percentage of patients (%) for whom there is a gap between practices and current recommendations regarding the choice of antibiotics, the daily dose and the number of doses per 24 hours, for the first episode of suspected or proven bacterial infection
Mean (SD) length of ICU stay (in days) from D0 (between beginning of antibiotics and cessation of antibiotics) | up to the end of hospitalization
  Mean (SD) length of ICU stay (in days) from D0
Mean (SD) length of hospital stay (in days) from D0 (between beginning of antibiotics and cessation of antibiotics) | up to the end of hospitalization
  Mean (SD) length of hospital stay (in days) from D0
All-cause hospital mortality rate (%) at D28 | up to 28 days
  All-cause hospital mortality is a mesure of all deaths, du to any cause, that occur in hospital during a clinical study.
Sepsis-related hospital mortality rate (%) at D28. | up to 28 days
  Sepsis-related hospitality mortality is a mesure of all deaths related to sepsis, that occur in hospital during a clinical study.
Percentage of patients with antibiotic-related adverse effects (%) (between beginning of antibiotics and cessation of antibiotics) | up to the end of hospitalization
  The antibiotic-related adverse effects are defined by a response to a drug which is noxious and unintended, and which occurs at doses normally used in man for the prophylaxis, diagnosis, or disease therapy, or for the modifications of physiological function (World Health Organization, 1972). They will be evaluated using Medical Dictionary for Regulatory Activities (MedDRA) coding, and severity and causality criteria. Only antibiotic-related adverse effects occurring in the same hospital stay as for the first episode will be taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Romain AMADIEU, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de TOULOUSE, Toulouse, France

REFERENCES:
- [Derived] Amadieu R, Brehin C, Chahine A, Grouteau E, Dubois D, Munzer C, Flumian C, Brissaud O, Ros B, Jean G, Brotelande C, Travert B, Savy N, Boeuf B, Ghostine G, Popov I, Duport P, Wolff R, Maurice L, Dauger S, Breinig S. Compliance with antibiotic therapy guidelines in french paediatric intensive care units: a multicentre observational study. BMC Infect Dis. 2024 Jun 12;24(1):582. doi: 10.1186/s12879-024-09472-0. PMID 38867164